CLINICAL TRIAL: NCT00894426
Title: Prospective, Observational, Multi-center, Non-interventional Study to Assess Patients Perception in SYmptoms Related to Morning Activity Based on Chronic Obstructive Lung Disease
Brief Title: Patient's Perception in Symptoms Related to Morning Activity Based on Chronic Obstructive Lung Disease
Acronym: SYMBOL
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: AstraZeneca, AstraZeneca
Other Study IDs: NIS-RKR-DUM-2009/1
Record Dates: First submitted 2009-04-28; First posted 2009-05-07 (Estimated); Last update posted 2010-12-03 (Estimated); Status verified 2010-12

CONDITIONS: COPD
Keywords: COPD; Symptom; Morning activity; Questionnaire
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- 1: Morning Symptoms (+)
- 2: Morning Symptoms (-)

SUMMARY:
The aim of this study is to assess the perception of chronic obstructive pulmonary disease (COPD) patients in symptoms related to morning activities. Also the researchers investigated how to describe the impact of symptoms on sleep quality and how to use the medication in Korea COPD treatments.

ELIGIBILITY:
Inclusion Criteria:

* COPD outpatients over 45 years old
* Lung function: post-FEV1 < 50%
* Current or ex-smoker > 10 packs per year
* Patients who were not on medication of ISC/FC at least 2 weeks

Exclusion Criteria:

* Ongoing exacerbation of COPD or within the previous 3 months
* History of asthma or allergic rhinitis
* Lung cancer or any other significant respiratory disease such as bronchiectasis, lung fibrosis, interstitial lung disease, tuberculosis, sarcoidosis
* Current participation in an interventional clinical trial

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The inclusion/exclusion criteria are designed to select subjects suffering from severe COPD (according to spirometric classification, GOLD stage III and IV) and in a stable state
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2009-05; Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
To assess the perception of COPD Patients in symptoms related to morning activities | At baseline and last visit (after 2~3 months)

SECONDARY OUTCOMES:
To assess the patient's perception of the variability of symptoms | At baseline and last visit (after 2~3 months)
To describe how patients use their COPD treatments | At baseline and last visit (after 2~3 months)
To investigate factors that may influence the patient's perception of symptom variability (such as patient characteristics, COPD treatments, co morbidities, etc…) | At baseline and last visit (after 2~3 months)

CONTACTS AND LOCATIONS:
Overall Officials: Joonwoo Bahn, Study Director — Astrazenca Korea, Medical Department
Locations (3):
- South Korea (3):
  - Research Site, Daegu
  - Research Site, Gyongiju
  - Research Site, Pohang